CLINICAL TRIAL: NCT03174158
Title: A Text Messaging Intervention for Smoking Cessation Among Community Health Center Patients
Brief Title: A Text Messaging Program for Smokers in Primary Care
Acronym: GR2Q
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Gina Kruse, Assistant Professor in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000960; 1K23DA038717-01A1 (NIH)
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Smoking Cessation
Keywords: text messaging
MeSH Terms: conditions — Smoking Cessation | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: 4 arm randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Brief advice (Active Comparator): Usual care plus brief telephone advice to quit tobacco delivered by a clinical research coordinator who underwent Tobacco Treatment Specialist core training.
  Interventions: Behavioral: Brief advice
- Text messaging (Experimental): Patients randomized to the text messaging program are offered a 12-week text messaging. The text messaging intervention will use content from the National Cancer Institute's SmokeFreeTXT library, content for smokers not ready to quit from SmokeFreeTXT and a pilot feasibility study conducted by the PI, and new messages supporting nicotine replacement medication adherence. The text messaging program will be personalized using subject's first name, the telephone number for the Massachusetts General Hospital (MGH) tobacco cessation counseling services and the Massachusetts state quitline. Smokers receiving the intervention will be sent from 0 and 5 text messages per day.
  Interventions: Behavioral: Text messaging; Behavioral: Brief advice
- Mailed nicotine replacement therapy (Experimental): Subjects randomized to mailed nicotine replacement therapy will be offered a 2 week supply of nicotine replacement therapy mailed to their home address. Daily smokers planning to quit in the next 30 days will be offered nicotine patches (14 or 21 mg patches) and lozenges (2 or 4 mg lozenges) dosed according to package instructions. Non-daily smokers planning to quit will be offered a 2 week allotment of 2 mg lozenges alone. Smokers not planning to quit will be offered one box of lozenges (72 count box of 4 mg or 2 mg lozenges based on time to first cigarette as above per package instructions) to use when they are not smoking during their practice quit attempt.
  Interventions: Drug: Mailed nicotine replacement therapy; Behavioral: Brief advice
- Text messaging + mailed NRT (Experimental): Subjects will be offered both the 12 week text message program and 2 weeks of mailed nicotine replacement therapy.
  Interventions: Drug: Mailed nicotine replacement therapy; Behavioral: Text messaging; Behavioral: Brief advice

INTERVENTIONS:
Drug: Mailed nicotine replacement therapy — Daily smokers will be offered patches and lozenges dosed according to package instructions (patches dosed according to cigarettes smoked per day and lozenges dosed according to time to first cigarette). Non-daily smokers will be offered a 2 week supply of 2 mg lozenges. Smokers not ready to quit will be offered one box of lozenges dosed according to time to first cigarette to use in a practice quit attempt.
  Arms: Mailed nicotine replacement therapy; Text messaging + mailed NRT
Behavioral: Text messaging — 12 week text messaging program tailored to readiness to quit and quit date. Program includes content encouraging NRT use. Content is personalized with user's name and Massachusetts General Hospital resources.
  Arms: Text messaging; Text messaging + mailed NRT
Behavioral: Brief advice — Brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training

SUMMARY:
This study is a four arm pilot randomized controlled trial testing the effect of a 12 week text messaging intervention and a mailed nicotine medication intervention, alone and in combination to a control condition consisting of brief behavioral advice and usual care.

Research Aim 1: To test, in a 4 arm pilot randomized controlled trial (N=50/group), the effect of a text messaging program and mailed nicotine replacement therapy on smoking outcomes and medication use.

Hypothesis 1: A text messaging intervention will increase the proportion of smokers making a quit attempt compared to smokers receiving no text messaging.

Hypothesis 2: A text messaging intervention will increase adherence to nicotine replacement therapy compared to subjects receiving only 2 weeks of nicotine replacement therapy.

Hypothesis 3: A text messaging intervention will increase the rate of biochemically confirmed past 7-day point prevalent tobacco abstinence at end of treatment compared to subjects receiving no text messaging intervention.

Hypothesis 4: A text messaging intervention will increase the number of days not smoking compared to subjects receiving no text messaging intervention.

Hypothesis 5: A text messaging intervention will decrease the number of cigarettes smoked per day compared to subjects receiving no text messaging intervention.

DETAILED DESCRIPTION:
Background: Fifteen percent of U.S. adults continue to smoke despite the availability of effective smoking cessation treatment and healthcare systems are positioned to address this deficiency. Text messaging is a widespread technology which shows promise as a way to reach smokers and to connect them with treatment. Tobacco cessation support delivered by text message increases abstinence among smokers interested in quitting in community- or school-based settings. This has led to the creation of text messaging programs by the National Cancer Institute, SmokeFreeTXT, and others. However, little is known about the feasibility of delivering smoking cessation support by text message for smokers engaged in healthcare systems. Integrating text messaging programs within healthcare systems has clear advantages. Documentation of smoking status is one of the Meaningful Use standards. This documentation enables healthcare systems to identify their population of smokers and proactively target them with health interventions outside of the busy office visit. Text messaging programs originating from the physicians' practice may also leverage the influence physicians have on smokers' motivation to quit.

Text messaging has been used in healthcare systems to effectively improve medication adherence in other conditions. Adherence to smoking cessation medications is at least modestly associated with cessation and measures of adherence to smoking cessation medications suggest overall low adherence to cessation medications outside of clinical trials. Offering free nicotine replacement therapy along with the medication adherence advice in a text messaging intervention will allow us to evaluate of the effect of adherence messages on medication use.

Study design A pilot randomized controlled trial of 206 smokers who receive care in Massachusetts General Hospital-affiliated primary care practices will compare the effect of delivering behavioral smoking cessation content with pharmacotherapy support by text message plus nicotine replacement therapy on self-reported quit attempts (intentional non-smoking for ≥24 hours), medication adherence, days not smoked, and smoking abstinence at the end of treatment. Smokers will be identified using the electronic health record, screened by their primary care provider, and proactively contacted by telephone by a clinical research coordinator. Potential subjects will be screened for eligibility by self-report and chart review by the Principal Investigator. Eligible subjects will be stratified by practice and readiness to quit (plan to quit smoking in the next 30 days vs no plan to quit smoking/plan to quit smoking in the next 6 months) and randomized 1:1:1:1 to 4 groups using a variable block randomization.

1. Brief advice (BA): Brief advice to quit smoking and usual care. Rationale: All subjects will receive brief advice from a trained clinical research coordinator. All primary care subjects also have access to guideline-concordant tobacco treatment through usual care with their primary care provider. Their primary care provider can refer them to in-person or telephone counseling and can prescribe medications.
2. Nicotine replacement therapy (NRT): Brief advice + 2 weeks of nicotine patches and/or lozenges mailed to subject. Rationale: In order to test the effect of text messaging on medication adherence, we need to have treatment groups receiving medication and medication plus text messaging. To deliver medication, mailed NRT, like text messaging, reaches patients outside of the busy office visit. Mailed NRT alone has also been shown to increase cessation and may itself be an effective intervention compared to brief advice and usual care.
3. Text messaging (TM): Brief advice + 12 week personalized, tailored text messaging program. Rationale: Text messaging shows promise as an intervention to help smokers to quit. However, it has not been well tested among primary care patients. Text messaging may connect those primary care smokers who do not access currently available treatment services like telephone counseling or prescribed medication with assistance outside of the clinic office.
4. Text messaging and nicotine replacement therapy (TM+NRT): Brief advice + 12 week personalized, tailored text messaging program + 2 weeks of nicotine patches and/or lozenges mailed to subject. Rationale: As above, in order to test the effect of text messaging on medication adherence, we need to have treatment groups receiving medication and medication plus text messaging. Text messaging has been shown to increase medication adherence in other conditions and medication adherence is suboptimal among users of smoking cessation medications. Integrating text messaging within healthcare systems offers opportunities to coordinate with pharmacotherapy and this 4 group design allows us to test the effect of text messaging alone on smoking outcomes and the effect of text messaging on NRT use.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Smoking status of current smoker in structured field of electronic health record (EHR)
* Language listed as English in EHR
* Massachusetts General Hospital patient, Partners healthcare primary care provider (PCP)
* PCP visit in the past 2 years
* Mobile telephone number listed in EHR

Exclusion Criteria:

* Not a current daily smoker defined as not having smoked ≥100 cigarettes in lifetime or self-report of less than daily current smoking
* Pregnant, planning to become pregnant in the next 3 months, or breastfeeding.
* Past 30-day use of nicotine replacement therapy, bupropion, or varenicline.
* Past 30-day use of Massachusetts state quit-line, "QuitWorks" or SmokefreeTXT programs
* Prior serious adverse reaction to the nicotine patch or lozenge defined as any reaction that was life-threatening, required hospitalization, or other clinical evaluation
* Ever had an allergy to nicotine patch
* Weight < 100 pounds
* Unstable coronary disease
* Unstable arrhythmia
* Dementia or active psychosis or schizoaffective disorder affecting ability to consent
* Willing and able to receive and participate with a text message program for up to 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina R Kruse, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massacusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kruse GR, Park ER, Chang Y, Haberer JE, Abroms LC, Shahid NN, Howard S, Haas JS, Rigotti NA. Proactively Offered Text Messages and Mailed Nicotine Replacement Therapy for Smokers in Primary Care Practices: A Pilot Randomized Trial. Nicotine Tob Res. 2020 Aug 24;22(9):1509-1514. doi: 10.1093/ntr/ntaa050. PMID 32198520
- [Derived] Kruse GR, Park E, Haberer JE, Abroms L, Shahid NN, Howard SE, Chang Y, Haas JS, Rigotti NA. Proactive text messaging (GetReady2Quit) and nicotine replacement therapy to promote smoking cessation among smokers in primary care: A pilot randomized trial protocol. Contemp Clin Trials. 2019 May;80:48-54. doi: 10.1016/j.cct.2019.03.006. Epub 2019 Mar 25. PMID 30923022

RESULTS

PARTICIPANT FLOW:
Groups:
- Text Messaging: Text messaging: 12 week text messaging program tailored to readiness to quit and quit date. Program includes content encouraging NRT use. Content is personalized with user's name and Massachusetts General Hospital resources.
  Brief advice: Brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist training
- Mailed Nicotine Replacement Therapy: Mailed nicotine replacement therapy: Daily smokers will be offered patches and lozenges dosed according to package instructions (patches dosed according to cigarettes smoked per day and lozenges dosed according to time to first cigarette). Non-daily smokers will be offered a 2 week supply of lozenges.
  Brief advice: Brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist training
- Text Messaging + Mailed NRT: Mailed nicotine replacement therapy: Daily smokers will be offered patches and lozenges dosed according to package instructions (patches dosed according to cigarettes smoked per day and lozenges dosed according to time to first cigarette). Non-daily smokers will be offered a 2 week supply of lozenges.
  Text messaging: 12 week text messaging program tailored to readiness to quit and quit date. Program includes content encouraging NRT use. Content is personalized with user's name and Massachusetts General Hospital resources.
  Brief advice: Brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist training
Period: Overall Study
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Started | 39 | 39 | 36 | 39
Completed | 35 | 37 | 34 | 38
Not Completed | 4 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT | Total
Number analyzed (Participants) | 39 | 39 | 36 | 39 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.8) | 54.0 (12.5) | 52.6 (9.1) | 51.5 (11.1) | 53.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 23 | 21 | 87
  Male | 18 | 17 | 13 | 18 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 34 | 27 | 24 | 31 | 116
  Black, non-Hispanic | 2 | 3 | 8 | 4 | 17
  Hispanic | 2 | 5 | 1 | 4 | 12
  Mixed race | 0 | 3 | 3 | 0 | 6
  Other | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 36 | 39 | 153
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 15.5 (7.1) | 13.6 (7.7) | 16.6 (6.8) | 15.4 (6.5) | 15.3 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Quit Attempts
Description: Self-reported quit attempt in the last 12 weeks defined as intentional not smoking for 24 hours or more ("During the past 12 weeks, have you quit smoking intentionally for 1 day or longer").
Time Frame: End of treatment (12 week post-enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 39 | 39 | 36 | 39
Participants | 26 | 33 | 29 | 31
Statistical Analysis 1: Comparison: Brief Advice vs Text Messaging; Test type: Superiority; p = 0.07, Chi-squared — a priori p value threshold < 0.05
Statistical Analysis 2: Comparison: Brief Advice vs Mailed Nicotine Replacement Therapy; Test type: Superiority; p = 0.18, Chi-squared; a priori threshold p<0.05
Statistical Analysis 3: Comparison: Brief Advice vs Text Messaging + Mailed NRT; Test type: Superiority; p = 0.21, Chi-squared — a priori threshold p<0.05

2. Secondary Outcome: 7 Day Point Prevalent Abstinence
Description: Self-reported abstinence "Have you smoked, even a puff, in the past 7 days?"
Time Frame: 6 weeks post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 39 | 39 | 36 | 39
Participants | 4 | 7 | 7 | 8

3. Secondary Outcome: 7 Day Point Prevalent Abstinence
Description: Self-reported abstinence "Have you smoked, even a puff, in the past 7 days?"
Time Frame: 12 weeks post-enrollment (end of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 39 | 39 | 36 | 39
Participants | 4 | 10 | 10 | 9

4. Secondary Outcome: Milligrams of Nicotine Medication Used
Description: Self-reported milligrams of nicotine medication used
Time Frame: week 2 post enrollment
Measure: Mean (Standard Deviation); unit: milligrams during week 2
Arm/Group | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 33 | 34
milligrams during week 2 | 84.2 (81.2) | 58.0 (91.3)

5. Secondary Outcome: Percentage of Days Not Smoked
Description: Self-reported, "In the past 30 days, how many days did you have at least one cigarette?"
Time Frame: 12 weeks post-enrollment (end of treatment)
Measure: Mean (Standard Deviation); unit: percentage of past 30 days
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 37 | 38 | 35 | 38
percentage of past 30 days | 23.7 (32.2) | 37.2 (32.0) | 29.0 (32.1) | 36.1 (35.5)

6. Secondary Outcome: Exhaled Carbon Monoxide
Description: Exhaled carbon monoxide measured among self-reported quitters less than or equal to 9 parts per million
Time Frame: 12 weeks post-enrollment (end of treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Mailed Nicotine Replacement Therapy: Mailed nicotine replacement therapy: Daily smokers will be offered patches and lozenges dosed according to package instructions (patches dosed according to cigarettes smoked per day and lozenges dosed according to time to first cigarette). Non-daily smokers will be offered a 2 week supply of lozenges.
  Brief advice: Brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training
- Text Messaging + Mailed NRT: Mailed nicotine replacement therapy: Daily smokers will be offered patches and lozenges dosed according to package instructions (patches dosed according to cigarettes smoked per day and lozenges dosed according to time to first cigarette). Non-daily smokers will be offered a 2 week supply of lozenges
  Text messaging: 12 week text messaging program tailored to readiness to quit and quit date. Program includes content encouraging NRT use. Content is personalized with user's name and Massachusetts General Hospital resources.
  Brief advice: Brief advice delivered by telephone by a clinical research coordinator who underwent Tobacco Treatment Specialist core training
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 1 | 3 | 3 | 2
Participants | 1 | 3 | 3 | 2

7. Secondary Outcome: Days Nicotine Medication Used
Description: Self-reported number of days nicotine lozenge and/or patch used
Time Frame: Total reported over 2 weeks post-enrollment
Measure: Mean (Standard Deviation); unit: days out of 2 weeks
Arm/Group | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 29 | 33
days out of 2 weeks | 5.3 (4.4) | 3.3 (4.3)

8. Secondary Outcome: Milligrams Nicotine Medication Used
Description: Self-reported number of milligrams nicotine medication used
Time Frame: Total reported over 1 week post-enrollment
Measure: Mean (Standard Deviation); unit: milligrams during week 1
Arm/Group | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 30 | 36
milligrams during week 1 | 33.8 (54.8) | 22.3 (45.8)

9. Secondary Outcome: Change in Cigarettes Per Day
Description: Self-reported number of cigarettes per day on days smoked, change
Time Frame: 12 weeks post enrollment (end of treatment)
Measure: Mean (Standard Deviation); unit: change in cigarettes per day
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
Number analyzed (Participants) | 27 | 31 | 29 | 30
change in cigarettes per day | -9.3 (8.3) | -8.6 (6.7) | -11.3 (7.3) | -8.9 (6.9)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse event data was collected at each outcome assessment
Arm/Group | Brief Advice | Text Messaging | Mailed Nicotine Replacement Therapy | Text Messaging + Mailed NRT
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/36 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/36 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 14/36 | 7/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief Advice (N=39) | Text Messaging (N=39) | Mailed Nicotine Replacement Therapy (N=36) | Text Messaging + Mailed NRT (N=39)
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Anxiety or agitation (Psychiatric disorders) | 0 | 0 | 2 | 3
mouth soreness (General disorders) | 0 | 0 | 2 | 0
sleep disturbance (Psychiatric disorders) | 0 | 0 | 1 | 1
lightheadedness (General disorders) | 0 | 0 | 1 | 0
skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
bloating (Gastrointestinal disorders) | 0 | 0 | 1 | 0
headache (Nervous system disorders) | 0 | 0 | 1 | 0
(General disorders) | 0 | 0 | 2 | 0 — Patient reported general side effect, not specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT03174158/Prot_SAP_000.pdf